CLINICAL TRIAL: NCT06584565
Title: A Multicenter Study Based on Multi-omics Analysis to Predict the Early Prognosis and Recurrence Risk of Acute Ischemic Stroke
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-150
Record Dates: First submitted 2024-08-26; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Ischemic Stroke, Acute
Keywords: Stroke recurrence; Post-stroke cognitive impairment; Post-stroke depression
MeSH Terms: conditions — Ischemic Stroke | interventions — Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- modeling queue: The modeling queue is used to manage and prioritize tasks related to the development and training of models.
  Interventions: Other: microbiome; metabolomics; proteomics
- validation queue: The validation queue is designed to handle tasks related to the evaluation and validation of models.
  Interventions: Other: microbiome; metabolomics; proteomics

INTERVENTIONS:
Other: microbiome; metabolomics; proteomics — post-stroke change of microbiome; metabolomics; proteomics

SUMMARY:
Through a multicenter prospective AIS cohort study, we analyze the potential association of human proteome, microbiome and metabolome alterations with AIS prognosis, searching for key proteins, differential organisms and metabolites, combining experimental data at multiple molecular levels with computational models, and establishing early prediction models through machine learning-based prediction algorithms. While closely tracking the recurrence of stroke in AIS patients, we evaluate the predictive value of human proteome, microbiome and metabolites for stroke recurrence through a nested case-control study, which provides key reference information for exploring the unknown residual risk of AIS recurrence.

DETAILED DESCRIPTION:
Currently, the burden of brain vascular disease in China is the highest in the world, and among them, the incidence rate of acute ischemic stroke (AIS) is high, the recurrence rate is high, the disability rate is high, the mortality rate is high, and the social burden is heavy. With the increasing number of AIS patients, how to effectively prevent and treat them is a huge challenge facing us. The occurrence and development of AIS are caused by the joint action of multiple risk factors and mutual influence, and single technical means are difficult to deeply explore its complex mechanism. Therefore, building a risk prediction model for poor prognosis and recurrence based on multi-omics technology and layering risk factors for patients are the important research directions for the future. This study aims to establish a multi-center cohort by collecting fecal and blood samples from AIS patients and conducting proteomic, microbial and metabolomic detection. It records the prognosis and recurrence events and uses cross-omics analysis technology to explore the multi-omics network molecular mechanism and screen for new intervention targets. It establishes an early prediction model and explores the stroke secondary prevention strategy based on multi-omics data.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of AIS according to the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2018
2. Aged 18 to 75 years old
3. Stroke within 7 days of onset
4. Sign informed consent, provide relevant medical history information and provide biological specimens

Exclusion Criteria:

1. Severe impairment of consciousness (awareness score of NIHSS>1)
2. History of stroke within 12 months
3. Severe systemic disease including malignancy
4. ALT or AST> 2 times the upper limit of normal or severe liver disease
5. creatinine > 1.5 times the upper limit of normal or severe kidney disease
6. History of long-term drinking, drug use, and chemical poisoning (e.g., pesticide poisoning); Note: Long-term alcohol consumption, usually more than 5 years, over 40 g/day of alcohol for men and 20 g/day for women, or a history of heavy alcohol consumption within 2 weeks, over 80 g/day of alcohol
7. History of intestinal tumors, irritable bowel syndrome or inflammatory bowel disease or confirmed in the hospital
8. Unable to collect a stool specimen within 4 days of admission
9. Assessed to be unsuitable for participation in this study by the investigator

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population mainly includes patients who meet the diagnostic criteria for acute ischemic stroke (AIS), are aged between 18 and 75 years, have a stroke onset within the past 7 days, and have clear consciousness. Patients with severe systemic diseases, a recent history of stroke, severe liver or kidney disease, a history of long-term alcohol consumption, those unable to provide a sample, or those assessed by the investigator as unsuitable for participation in the study are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of new cardiovascular events and death | within 12 months after onset
  any stroke /TIA/ myocardial infarction/Vascular death

SECONDARY OUTCOMES:
Brain Injury Conditions | 3, 12 months after ischemic stroke
  Clinical investigators evaluate brain injury conditions according to head CT or MR, which including the signs of infarct lesions, hemorrhagic transformation post-infarction or cerebral edema.
Small Vessel Disease Burden | 3, 12 months after ischemic stroke
  Clinical investigators evaluate small vessel disease burden according to head CT or MR, which including the signs of white matter degeneration, lacunar infarctions, cerebral microbleeds or enlarged perivascular spaces.
Cerebrovascular Pathology | 3, 12 months after ischemic stroke
  Clinical investigators evaluate cerebrovascular pathology according to head CT or MR, which including the signs of vascular stenosis, vascular dissection or collateral circulation compensation.
Modified Rankin Scale ( mRS ) score | 7 day and 3, 12 months after ischemic stroke
  The MRS score is primarily used to measure the degree of disability and daily living ability of patients. The MRS score ranges from 0 to 6, with a total of 7 levels. The higher the score, the more severe the disability and the worse the prognosis.
National Institutes of Health Stroke Scale ( NIHSS ) score | 7 day and 3, 12 months after ischemic stroke
  The NIHSS score is commonly used to assess the degree of neurological impairment in patients with acute stroke. The NIHSS consists of 11 items, with a total score ranging from 0 to 42. Each item has different scoring criteria, typically ranging from 0 (normal) to 4 (most severe).
Activity of Daily Living Scale ( ADL ) score | 7 day and 3, 12 months after ischemic stroke
  The ADL score is primarily used to measure a person's ability to perform basic daily activities. This study uses the Barthel Index scoring method, which ranges from 0 to 100 points, with scoring items including eating, bathing, grooming, dressing, bowel control, bladder control, toileting, transferring, mobility and stairs. A higher score indicates greater independence, while a lower score indicates greater dependence.
Mini-mental State Examination ( MMSE ) score | 3, 12 months after ischemic stroke
  The MMSE (Mini-Mental State Examination) is a tool used to assess cognitive function, including orientation, memory, attention, language skills, calculation ability, and visuospatial skills. It is commonly used to screen for dementia in older adults. The MMSE has a total score of 30 points: a score of 24-30 suggests normal cognitive function, 18-23 indicates mild cognitive impairment, and 0-17 indicates moderate to severe cognitive impairment.
Montreal Cognitive Assessment ( MOCA ) score | 3, 12 months after ischemic stroke
  The MoCA is a tool used to assess cognitive impairment. Compared to the MMSE, the MoCA is more sensitive, particularly for detecting mild cognitive impairment (MCI). The MoCA has a total score of 30 points: a score of 26-30 suggests normal cognitive function, 18-25 indicates mild cognitive impairment (MCI), and 0-17 indicates moderate to severe cognitive impairment. Typically, individuals with lower educational levels (less than 12 years of education) receive an additional point as an adjustment to their total score.
Hamilton Depression Scale ( HAMD ) score | 3, 12 months after ischemic stroke
  The HAMD is a clinical scale used to assess the severity of depression. This study uses the 17-item version (HAMD-17), which covers a range of symptoms, including mood, sleep, appetite, and somatic symptoms. The total score ranges from 0 to 52, with each item rated based on the severity of symptoms, typically from 0 (no symptoms) to 4 (severe symptoms).
Hamilton Anxiety Scale ( HAMA ) score | 3, 12 months after ischemic stroke
  The HAMA is a clinical scale used to assess the severity of anxiety symptoms. It consists of 14 items, each evaluating different symptoms related to anxiety. These symptoms cover both psychological and somatic manifestations of anxiety. Each item is rated based on the severity of symptoms, with scores ranging from 0 (no symptoms) to 4 (very severe symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital,Southern Medical University, Guangzhou, Guangdong, China